CLINICAL TRIAL: NCT01424644
Title: A Phase 4, Placebo-Controlled, Randomized Study to Evaluate the Immunogenicity and Safety of a Combined Tetanus, Reduced Diphtheria Toxoid, Acellular Pertussis Vaccine (Tdap, Boostrix®) and Quadrivalent Human Papillomavirus [Types 6, 11, 16, 18] Recombinant Vaccine (Gardasil®) in Healthy Adolescents When Administered With MenACWY Conjugate Vaccine
Brief Title: A Phase 4, Placebo-Controlled, Randomized Study to Evaluate the Immunogenicity and Safety of HPV and Tdap When Administered With MenACWY in Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V59_40; 2011-000476-34 (EudraCT Number)
Record Dates: First submitted 2011-08-23; First posted 2011-08-29 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Meningococcal Meningitis
Keywords: meningitis; human papillomavirus; tetanus; diptheria; pertussis
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis; Tetanus; Whooping Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo + Tdap + HPV (Placebo Comparator): This group will receive Tdap, HPV and placebo concomitantly for the first vaccination. The second and third doses of HPV vaccine will be administered to all subjects 2 and 6 months after the first dose. All subjects will have serum samples collected at Visit 1 (baseline), Visit 2 (31 days) and Visit 5 (7 months after visit 1) for serology testing.
  Interventions: Biological: Placebo + Combined Tetanus, Reduced Diphtheria Toxoid, Acellular Pertussis Vaccine + Quadrivalent Human Papillomavirus Vaccine
- MenACWY-CRM + Tdap + HPV (Experimental): This group will receive Tdap, HPV and MenACWY-CRM concomitantly. The second and third doses of HPV vaccine will be administered to this group 2 and 6 months after the first dose. All subjects will have serum samples collected at Visit 1 (baseline), Visit 2 (31 days) and Visit 5 (7 months after visit 1) for serology testing.
  Interventions: Biological: MenACWY-CRM Conjugate Vaccine + Combined Tetanus, Reduced Diphtheria Toxoid, Acellular Pertussis Vaccine + Quadrivalent Human Papillomavirus Vaccine

INTERVENTIONS:
Biological: Placebo + Combined Tetanus, Reduced Diphtheria Toxoid, Acellular Pertussis Vaccine + Quadrivalent Human Papillomavirus Vaccine — All three vaccines were administered concomitantly. Quadrivalent Human Papillomavirus [Types 6, 11, 16, 18] Recombinant Vaccine is GARDASIL®.
  Reduced Diphtheria Toxoid, Acellular Pertussis Vaccine(Tdap) is Boostrix®.
  Arms: Placebo + Tdap + HPV
Biological: MenACWY-CRM Conjugate Vaccine + Combined Tetanus, Reduced Diphtheria Toxoid, Acellular Pertussis Vaccine + Quadrivalent Human Papillomavirus Vaccine — All three vaccines were administered concomitantly. MenACWY-CRM contains diphtheria-like toxoid as carrier for the capsular polysaccharides. Quadrivalent Human Papillomavirus [Types 6, 11, 16, 18] Recombinant Vaccine is GARDASIL®.
  Reduced Diphtheria Toxoid,Acellular Pertussis Vaccine(Tdap) is Boostrix®.
  Arms: MenACWY-CRM + Tdap + HPV

SUMMARY:
The main objective is to determine whether immune responses to Tdap (GlaxoSmithKline, Boostrix®) and HPV vaccine (Merck & Co., Inc., Gardasil®) when administered concomitantly with MenACWY are comparable to responses elicited by these vaccines when given alone.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for enrollment in this study were female and male individuals who had been shown to be healthy and who were:

1. 11-18 years of age inclusive who had given their written consent/assent and if applicable, whose parents or legal guardians had given written informed consent at the time of enrollment;

   * Available for all visits and telephone calls scheduled for the study;
   * In good health as determined by:

     * Medical history
     * Physical assessment
     * Clinical judgment of the investigator
2. Had been properly vaccinated against diphtheria, tetanus, and pertussis per local regulations;
3. Subjects who were current with childhood DTP-containing vaccinations per local guidelines. Any previous vaccinations containing DTP must have been received at least 5 years before study enrollment and no prior adolescent vaccinations (11-18 years of age) containing DTP vaccines were allowed.
4. For female subjects, who had a negative urine pregnancy test.
5. Any female subject who is sexually active committed to practice appropriate birth control.

Exclusion Criteria:

Individuals not eligible to be enrolled in the study were those:

1. Who were unwilling to give their written assent / consent
2. Who were breastfeeding
3. Who was, and/or whose parents or legal guardians were perceived to be unreliable or unavailable for the duration of the study period
4. Who had previous confirmed or suspected disease caused by N. meningitidis
5. Who had household contact with and/or intimate exposure to an individual with culture-proven N. meningitidis infection within 60 days prior to enrollment
6. Who had previously been immunized with a meningococcal vaccine or vaccine containing meningococcal antigen(s) (licensed or investigational). (Exception: Receipt of OMP-containing Hib vaccines was permitted)
7. Who had received prior human papillomavirus (HPV) vaccine
8. Who had received investigational agents or vaccines within 30 days prior to enrollment or who expected to receive an investigational agent or vaccine prior to completion of the study
9. Who had received live licensed vaccines within 30 days and inactive vaccine within 15 days prior to enrollment or for whom receipt of a licensed vaccine is anticipated during the study period.

   (Exception: Influenza vaccine could be administered up to 15 days prior to each study immunization and no less than 15 days after each study vaccination)
10. Who had experienced, within the 7 days prior to enrollment, significant acute or chronic infection (for example requiring systemic antibiotic treatment or antiviral therapy) or had experienced fever (defined as body temperature ≥ 38°C) within 3 days prior to enrollment
11. Who had any serious acute, chronic or progressive disease such as

    * History of cancer
    * Complicated diabetes mellitus
    * Advanced arteriosclerotic disease
    * Autoimmune disease
    * HIV infection or AIDS
    * Blood dyscrasias
    * Congestive heart failure
    * Renal failure
    * Severe malnutrition (Note: Subjects with mild asthma were eligible for enrollment. Subjects with moderate or severe asthma requiring routine use of inhaled or systemic corticosteroids were not eligible for enrollment)
12. Who had epilepsy, any progressive neurological disease or history of Guillain-Barre syndrome
13. Who had a history of anaphylaxis, serious vaccine reactions, or allergy to any vaccine component, including latex allergy
14. Who had a known or suspected impairment/alteration of immune function, either congenital or acquired or resulting from (for example):

    * Receipt of immunosuppressive therapy within 30 days prior to enrollment (systemic corticosteroids administered for more than 5 days, or in a daily dose > 1 mg/kg/day prednisone or equivalent during any of 30 days prior to enrollment, or cancer chemotherapy)
    * Receipt of immunostimulants
    * Receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 90 days prior to enrollment and for the full length of the study
15. Who were known to have a bleeding diathesis, or any condition that may be associated with a prolonged bleeding time;
16. Who have Down's syndrome or other known cytogenic disorders;
17. Who and/or whose families were planning to leave the area of the study site before the end of the study period;
18. Who had any condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
19. Who were relatives of the study personnel.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 801 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (20):
- United States (17):
  - Birmingham Pediatrics, 806 Saint Vincent's Drive, Suite 615, Birmingham, Alabama
  - Prairie Fields Family Medicine, 350 W. 23rd Street, Suite A, Fremont, California
  - Madera Family Medical Group, 1111 W. Fourth Street, Madera, California
  - Clinical Research Advantage / Colorado Springs Health Partners, 6340 Barnes Road, Colorado Springs, Colorado
  - Dayton Clinical Research, 1100 Salem Ave, Dayton, Florida
  - Altamonte Pediatric Associates, 101 N. Country Club Rd. #113, Lake Mary, Florida
  - Pediatrics and Adolescent Medicine, 2155 Post Oak Tritt Road, Suite 100, Marietta, Georgia
  - Clinical Research Advantage / Ridge Family Physicians, 201 Ridge Street, Suite 201, Council Bluffs, Iowa
  - Columbia Medical Practice, 5450 Knoll North Drive, Suite 215, Columbia, Maryland
  - Roslindale Pediatrics Associates, 1153 Centre Street, Suite 31, Boston, Massachusetts
  - Bellevue Family Practice, 2206 Longo Suite 201, Bellevue, Nebraska
  - Complete Children's Health, 8201 Northwoods Drive, Lincoln, Nebraska
  - Meridian Clinical Research, 3319 North, 107th Street, Omaha, Nebraska
  - Pediatrics and Adolescent Medicine, 120 Stonebridge Parkway, Suite 410, Woodstock, New York
  - Capitol Pediatrics and Adolescent Center, 3801 Computer Drive Suite 200, Raleigh, North Carolina
  - Ohio Pediatric Research Association, 7371 Brandt Pike Suite C, Huber Heights, Ohio
  - Omega Medical Research, 400 Bald Hill Road, Warwick, Rhode Island
- Italy (3):
  - HOSPITAL"SAN MARTINO". Department of Health Sciences University of Genoa, Via Pastore, 1, Genoa
  - Hospital "Maggiore della Carità". Pediatric Clinic, Corso Mazzini, 18, Novara
  - Hospital of Taranto- Unit of Hygiene and Publich Health Vaccination Center, Viale Magna Grecia, 173, Taranto

REFERENCES:
- [Derived] Miao Y, Mzolo T, Pellegrini M. Immunogenicity of a Quadrivalent Human Papillomavirus Vaccine When Co-Administered with Tetanus-Reduced Diphtheria-Acellular Pertussis and Quadrivalent Meningococcal Conjugate Vaccines in Healthy Adolescents: Results from a Randomized, Observer-Blind, Controlled Trial. Infect Dis Ther. 2019 Sep;8(3):335-341. doi: 10.1007/s40121-019-00258-5. Epub 2019 Aug 3. PMID 31377946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in two countries (US and Italy).
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- MenACWY-CRM+Tdap+HPV: Subjects received one dose of Tdap, MenACWY-CRM, and HPV concomitantly on day 1. A second and third dose of HPV was administered at 2 and 6 months, respectively, after the first dose.
- Placebo+Tdap+HPV: Subjects received one dose of Tdap, placebo, and HPV concomitantly on day 1. A second and third dose of HPV was administered at 2 and 6 months, respectively, after the first dose.
Period: Overall Study
Arm/Group | MenACWY-CRM+Tdap+HPV | Placebo+Tdap+HPV
Started | 402 | 399
Completed | 369 | 372
Not Completed | 33 | 27
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 9 | 12
Not completed — Lost to Follow-up | 16 | 12
Not completed — Protocol Violation | 4 | 3
Not completed — Administrative Reason | 1 | 0
Not completed — Unable to Classify | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM+Tdap+HPV | Placebo+Tdap+HPV | Total
Number analyzed (Participants) | 402 | 399 | 801
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (1.7) | 11.8 (1.5) | 11.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 155 | 324
  Male | 233 | 244 | 477

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Anti-diphtheria and Anti-tetanus Antibody Concentrations ≥ 0.1 IU/mL When Tdap is Administered Concomitantly With HPV and MenACWY-CRM Vaccine Compared to Tdap Given Concomitantly With HPV and Placebo
Description: The percentages of subjects with anti-diphtheria and anti-tetanus antibody concentrations ≥ 0.1 IU/mL (as measured by ELISA) following concomitant administration of Tdap with HPV and MenACWY-CRM vaccine as compared to concomitant administration of Tdap with HPV and placebo.
Time Frame: 1 month post Tdap vaccination.
Population: Analysis was done on the Tdap per-protocol population, i.e., all subjects who received all the relevant doses of vaccine correctly, and provided serology results at one month postvaccination, and had no major protocol violation as defined prior to unblinding.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM+Tdap+HPV | Placebo+Tdap+HPV
Number analyzed (Participants) | 376 | 382
percentages of subjects
  Day 1 (diphtheria) (N=375, 380) | 5 [3 to 8] | 3 [2 to 5]
  One month post dose (diphtheria) | 95 [93 to 97] | 82 [78 to 86]
  Day 1 (tetanus ) (N=375, 380) | 28 [24 to 33] | 28 [23 to 32]
  One month post dose (tetanus ) | 99 [97 to 100] | 98 [97 to 99]
Statistical Analysis 1: Comparison: MenACWY-CRM+Tdap+HPV vs Placebo+Tdap+HPV; Non-inferiority of anti-diphtheria immune response following concomitant administration of Tdap with HPV and MenACWY-CRM as compared to concomitant administration of Tdap with HPV and placebo; Test type: Non-Inferiority or Equivalence — The immune response to diphtheria toxin for the MenACWY-CRM+Tdap+HPV group was considered non-inferior to that of the Placebo+Tdap+HPV group if the lower limit of the two-sided 95% CI of the difference in seroprotection rates [(MenACWY-CRM+Tdap+HPV) minus (Placebo+Tdap + HPV)] was greater than -10%, at 1 month after Tdap vaccination; Miettinen and Nurminen; Vaccine group difference = 13, 95% CI 2-sided [9 to 17]
Statistical Analysis 2: Comparison: MenACWY-CRM+Tdap+HPV vs Placebo+Tdap+HPV; Non-inferiority of anti-tetanus immune response following concomitant administration of Tdap with HPV and MenACWY-CRM as compared to concomitant administration of Tdap with HPV and placebo; Test type: Non-Inferiority or Equivalence — The immune response to tetanus toxin for the MenACWY-CRM+Tdap+HPV group was considered non-inferior to that of Placebo+Tdap+HPV group if the lower limit of the two-sided 95% CI of the difference in seroprotection rates [(MenACWY-CRM+ Tdap+HPV) minus (Placebo+Tdap + HPV)] was greater than -10%, at 1 month after Tdap vaccination; Miettinen and Nurminen; Vaccine group difference = 0, 95% CI 2-sided [-2 to 2]

2. Primary Outcome: Geometric Mean Concentrations of Antibodies Against Pertussis Antigens After Concomitant Administration of Tdap With HPV and MenACWY-CRM Compared to Concomitant Administration of Tdap With HPV and Placebo
Description: The geometric mean concentrations (GMCs) of antibodies against pertussis antigens (PT, FHA and PRN), as measured by ELISA, following concomitant administration of Tdap with HPV and MenACWY-CRM as compared to concomitant administration of Tdap with HPV and placebo.
Time Frame: 1 month post Tdap vaccination.
Population: Analysis was done on the Tdap per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | MenACWY-CRM+Tdap+HPV | Placebo+Tdap+HPV
Number analyzed (Participants) | 376 | 382
EU/mL
  PT (Day 1) (N= 375, 380) | 4.77 [4.11 to 5.53] | 4.16 [3.59 to 4.82]
  PT(One month post dose) | 44 [40 to 48] | 44 [40 to 48]
  FHA (Day 1) (N= 375, 380) | 24 [21 to 27] | 21 [18 to 23]
  FHA (One month post dose) | 202 [187 to 218] | 240 [222 to 259]
  PRN (Day 1) (N= 375, 380) | 20 [18 to 23] | 21 [18 to 24]
  PRN (One month post dose) | 330 [300 to 363] | 403 [367 to 443]
Statistical Analysis 1: Comparison: MenACWY-CRM+Tdap+HPV vs Placebo+Tdap+HPV; Non-inferiority of anti-PT immune response following concomitant administration of Tdap with HPV and MenACWY-CRM as compared to concomitant administration of Tdap with HPV and placebo; Test type: Non-Inferiority or Equivalence — The immune response to PT antigen for the MenACWY-CRM+Tdap+HPV group was considered non-inferior to that of the Placebo+Tdap+HPV group if the lower limit of the two-sided 95% CI of the ratio of the GMCs of the MenACWY-CRM +Tdap+HPV group to the Placebo+Tdap + HPV group was greater than 0.5, at 1 month after Tdap vaccination; ANOVA; Vaccine group ratio-Geometric mean conc = 1.01, 95% CI 2-sided [0.89 to 1.14]
Statistical Analysis 2: Comparison: MenACWY-CRM+Tdap+HPV vs Placebo+Tdap+HPV; Non-inferiority of anti-FHA immune response following concomitant administration of Tdap with HPV and MenACWY-CRM as compared to concomitant administration of Tdap with HPV and placebo; Test type: Non-Inferiority or Equivalence — The immune response to FHA antigen for the MenACWY-CRM+Tdap+HPV group was considered non-inferior to that of Placebo+Tdap+HPV group if the lower limit of the 95% CI of the difference [(MenACWY-CRM +Tdap+HPV) minus(Placebo+Tdap + HPV)] was greater than 0.5, at 1 month after Tdap vaccination; ANOVA; Vaccine group ratio- Geometric mean conc = 0.84, 95% CI 2-sided [0.76 to 0.93]
Statistical Analysis 3: Comparison: MenACWY-CRM+Tdap+HPV vs Placebo+Tdap+HPV; Non-inferiority of anti-PRN immune response following concomitant administration of Tdap with HPV and MenACWY-CRM as compared to concomitant administration of Tdap with HPV and placebo; Test type: Non-Inferiority or Equivalence — The immune response to PRN antigen for the MenACWY-CRM+Tdap+HPV group was considered non-inferior to that of Placebo+Tdap+HPV group if the lower limit of the 95% CI of the difference [(MenACWY-CRM+Tdap+HPV) minus(Placebo+Tdap + HPV)] was greater than 0.5, at 1 month after vaccination; ANOVA; Vaccine group ratio-Geometric mean conc = 0.82, 95% CI 2-sided [0.72 to 0.93]

3. Secondary Outcome: Geometric Mean hSBA Titers Against N. Meningitidis Serogroups A,C,W and Y at 1 Month After Men ACWY Vaccination.
Description: The immunogenicity was assessed in terms of geometric mean hSBA titers of MenACWY when administered concomitantly with Tdap and HPV at 1 month after 1 dose of MenACWY vaccination.
Time Frame: 1 month post MenACWY-CRM vaccination.
Population: Analysis was done on the MenACWY per-protocol population - all subjects who received all the relevant doses of vaccine correctly, and provided evaluable serum samples at baseline and one month postvaccination for at least one serogroup, and had no major protocol violation as defined prior to unblinding.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM+Tdap+HPV | Placebo+Tdap+HPV
Number analyzed (Participants) | 371 | 99
Titers
  Men A | 35 [29 to 42] | 2.13 [1.97 to 2.31]
  Men C (N=370, 97) | 59 [48 to 73] | 3.92 [3.3 to 4.66]
  Men W (N=369, 96) | 61 [53 to 69] | 12 [9.26 to 17]
  Men Y (N=369, 97) | 48 [40 to 58] | 3.54 [2.9 to 4.31]

4. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Adverse Events When Tdap and HPV Are Concomitantly Administered With MenACWY-CRM Compared to When Tdap and HPV Are Concomitantly Administered With Placebo
Description: The number of subjects reporting solicited local and systemic reactions following concomitant administration of MenACWY-CRM vaccine, Tdap and HPV vaccine as compared to concomitant administration of placebo with Tdap and HPV.
Time Frame: Day 1-7 after any vaccination.
Population: Analysis was done on solicited safety Set - All subjects in the exposed population who provided solicited AEs.
Measure: Number; unit: Subjects
Arm/Group | MenACWY-CRM+Tdap+HPV | Placebo+Tdap+HPV
Number analyzed (Participants) | 389 | 385
Subjects
  Local | 209 | 164
  Injection site pain | 158 | 134
  Injection site erythema | 65 | 25
  Injection site induration | 61 | 37
  Systemic | 205 | 179
  Chills | 60 | 50
  Nausea | 54 | 39
  Malaise | 57 | 44
  Myalgia | 115 | 101
  Arthralgia | 35 | 43
  Headache | 113 | 95
  Rash | 4 | 7
  Fever ≥ 38°C | 9 | 8
  Other | 88 | 80
  Stayed home due to reaction | 25 | 33
  Analgesic / Antipyretic medication used | 74 | 65

5. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events When Tdap and HPV Are Concomitantly Administered With MenACWY-CRM Compared to When Tdap and HPV Are Concomitantly Administered With Placebo
Description: The number of subjects reporting any unsolicited adverse reactions (AEs) when Tdap and HPV are concomitantly administered with MenACWY-CRM as compared to when Tdap and HPV vaccine are concomitantly administered with placebo.
  Note: A total of 2 MenACWY-CRM+Tdap+HPV subjects reported AEs leading to premature withdrawal - one subject due to treatment emergent AE and another subject prior to study vaccination on day 1.
Time Frame: Throughout the study (Day 1 to Day 211).
Population: Analysis was done on overall safety population - All subjects in the exposed population who provided postvaccination and post-baseline safety data.
Measure: Number; unit: Subjects
Arm/Group | MenACWY-CRM+Tdap+HPV | Placebo+Tdap+HPV
Number analyzed (Participants) | 396 | 397
Subjects
  Any AEs | 201 | 197
  At least possibly related AEs | 17 | 14
  Serious AEs | 4 | 3
  AEs leading to Premature Withdrawal | 2 | 0

ADVERSE EVENTS:
Time Frame: From day 1 through day 211.
Description: Serious adverse events (SAEs) were collected from Day 1 through Day 211.
  Note: Among 801 subjects in the enrolled population (reported in the participant flow module), 793 subjects were exposed to the study vaccines.
Arm/Group | MenACWY-CRM+Tdap+HPV | Placebo+Tdap+HPV
Serious Adverse Events (participants affected / at risk) | 4/396 | 3/397
Other Adverse Events (participants affected / at risk) | 288/396 | 248/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM+Tdap+HPV (N=396) | Placebo+Tdap+HPV (N=397)
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Type 1 Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM+Tdap+HPV (N=396) | Placebo+Tdap+HPV (N=397)
Nausea (Gastrointestinal disorders) | 59 | 42
Chills (General disorders) | 65 | 50
Injection site erythema (General disorders) | 79 | 30
Injection site induration (General disorders) | 69 | 43
Injection site pain (General disorders) | 193 | 165
Malaise (General disorders) | 59 | 45
Pharyngitis (Infections and infestations) | 22 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 47
Myalgia (Musculoskeletal and connective tissue disorders) | 117 | 109
Headache (Nervous system disorders) | 128 | 105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days